CLINICAL TRIAL: NCT04750057
Title: An Early Access Program for Anifrolumab Treatment in Adult Patients With Active Systemic Lupus Erythematosus - AMANA
Brief Title: Anifrolumab Early Access Program
Acronym: AMANA
Status: No longer available | Type: Expanded Access
Sponsor: AstraZeneca (Industry)
Collaborators: Clinigen, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00027
Record Dates: First submitted 2021-02-09; First posted 2021-02-11 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Anifrolumab — Multi-centre, open-label, early access program (EAP) designed to provide access to intravenous (IV) treatment regimen of 300 mg anifrolumab (MEDI-546) every 4 weeks (Q4W) for eligible patients with moderate-to-severe active SLE while receiving standard therapy.
  Other Names: MEDI-546, D3461

SUMMARY:
To provide early access (ie, before marketing authorisation) to anifrolumab 300 mg IV Q4W while receiving standard therapy in adult patients with moderate-to-severe active SLE

DETAILED DESCRIPTION:
This is a multi-centre, open-label, early access program (EAP) designed to provide treatment access to intravenous (IV) treatment regimen of 300 mg anifrolumab (MEDI-546) every 4 weeks (Q4W) for eligible patients with moderate-to-severe active SLE while receiving standard therapy. Anifrolumab will be provided free of charge to the patients entering this program.This global EAP will be opened in a sequential fashion, country by country, based on the requesting Treating Physician(s) and local regulations

ELIGIBILITY:
Population A:

Inclusion Criteria:

1. Received anifrolumab or placebo in the long-term extension study, D3461C00009, and are within 12 weeks of Week 164 (follow-up visit 2).
2. Provided written informed consent before any program-related procedures are performed.
3. Adequate peripheral venous access.
4. Females of childbearing potential must use two effective methods of avoiding pregnancy, only one of which is a barrier method, from screening until 12 weeks after final dose of anifrolumab, unless the patient is surgically sterile (eg, bilateral oophorectomy or complete hysterectomy), has a sterile male partner, is at least 1 year ostmenopausal, or practises sustained abstinence consistent with the patient's customary lifestyle. Postmenopausal is defined as at least 1 year since last menses and the patient has an elevated follicle-stimulating hormone (FSH) level greater than the local laboratory value of post-menopausal at screening - as detailed in Section 5.4.3.
5. All males (sterilised or non-sterilised) who are sexually active must use a condom (with spermicide where commercially available) from Day 1 (first dose of anifrolumab) until at least 12 weeks after receiving the final dose of anifrolumab. It is strongly recommended that the female partner of a male patient also uses an effective method of contraception (other than a barrier method) throughout this period. Male patients must not donate sperm while taking part in the EAP and for 12 weeks after their last dose of anifrolumab - see Section 5.4.3 for further details.
6. Females with an intact cervix must have a documented normal Pap smear without documented malignancy (eg, no signs of cervical intraepithelial neoplasia [CIN] grade III, carcinoma in situ [CIS] or adenocarcinoma in situ [AIS]) within 2 years of entering this EAP and receiving anifrolumab. Any abnormal Pap smear result documented within 2 years before receiving anifrolumab must be repeated to confirm patient eligibility.
7. COVID-19: Any negative polymerase chain reaction (PCR) test result (central laboratory) at screening and no known or suspected COVID-19 exposure within 2 weeks prior to screening. If there is a known or suspected exposure, a patient must be negative upon retest obtained after 2 weeks and must remain asymptomatic for inclusion in the study. Note: Patients positive at screening may be re-screened after 3 months provided there has been no development of severe COVID-19 disease or sequalae.

Exclusion Criteria:

1. Discontinued anifrolumab or placebo, for any reason including an AE, before completing Year 3 of the treatment period for study 09 or study 1145.
2. Major medical event, such as cerebrovascular accident (CVA), myocardial infarction (MI), malignancy, opportunistic infection, suicide attempt, or that, in the opinion of the Treating Physician, would interfere with patient safety.
3. Any other condition that, in the opinion of the Treating Physician, would interfere with patient safety.
4. Active severe or unstable neuropsychiatric SLE where, in the opinion of the Treating Physician, protocol-specified standard therapy is insufficient and utilisation of a more aggressive therapeutic approach, such as adding IV cyclophosphamide and/or high dose IV pulse corticosteroid therapy or other treatments not permitted in the protocol, is indicated.
5. Active severe SLE-driven renal disease where, in the opinion of the Treating. Physician or delegate, protocol-specified standard therapy is insufficient and utilisation of a more aggressive therapeutic approach, such as adding IV cyclophosphamide and/or high dose IV pulse corticosteroid therapy or other treatments not permitted in the protocol, is indicated.
6. Is receiving any of the following medications:

   1. Azathioprine > 200 mg/day
   2. Mycophenolate mofetil > 2 g/day or mycophenolic acid > 1.44 g/day
   3. Oral, subcutaneous (SC), or intramuscular (IM) methotrexate > 25 mg/week
   4. Oral prednisone > 40 mg/day (or prednisone equivalent - see Appendix E1)
   5. Mizoribine > 150 mg/day
   6. Biologics eg, belimumab, rituximab
7. Received any of the following:

   1. Live or attenuated vaccine within 8 weeks before signing the ICF. Note: administration of inactivated vaccines is acceptable - the Sponsor recommends that Treating Physicians ensure all patients are up to date on required vaccinations, including influenza (inactivated/recombinant) before EAP entry.
   2. Restricted medications listed in Appendix D if the washout period is not met.
8. Received any investigational product (small molecule or biologic agent) within 4 weeks or 5 half-lives (whichever is greater) before signing the ICF (see Appendix D).
9. Received any commercially available biologic agent within 5 half-lives before signing ICF (see Appendix D).
10. Received B-cell-depleting therapy (including, but not limited to: ocrelizumab, ofatumumab, atacicept, obinutuzumab, rituximab) within 26 weeks before signing the ICF; within 40 weeks for atacicept (see Appendix D) or if therapy was administered 26 weeks or more ago (40 weeks for atacicept), absolute B-cell count should not be less than the lower limit of normal (LLN) or baseline (whichever is lower) before receipt of B-cell-depleting therapy.
11. Positive hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
12. Known history of allergy or reaction to any component of anifrolumab or history of anaphylaxis to any human gamma globulin therapy.
13. COVID-19: Any history of severe COVID-19 infection (e.g. requiring hospitalisation, intensive care unit (ICU) care or assisted ventilation) or any prior COVID-19 infection with unresolved sequelae. Any acute COVID-19 infection (laboratory confirmed or suspected based on clinical symptoms) within the last 3 months prior to screening.

Population B:

Inclusion criteria:

1. Patients who have:

   1. Completed study D3461C0009 safety follow-up period (Week 164), and more than 12 weeks since Week 164 (safety follow-up visit 2); OR
   2. Completed safety follow-up period in phase 2 study CD1145; OR
   3. Not previously taken part in any anifrolumab clinical study and have attempted the standard therapeutic options at the maximum tolerated dose (see inclusion criterion 2); AND

   i. Are not eligible for enrollment in an anifrolumab clinical study, AND ii. Have moderate to severe SLE (no lupus nephritis or severe CNS lupus)
2. Attempted standard therapies, such as an antimalarial, therapeutic doses of oral corticosteroids, minimum of 2 immunosuppressants and biologics (belimumab or rituximab, if available in their country) from the following therapeutic options at the maximum tolerated dose:

   1. Azathioprine ≤ 200 mg/day
   2. Antimalarial (eg, chloroquine, hydroxychloroquine, quinacrine)
   3. Mycophenolate mofetil ≤ 2 g/day or mycophenolic acid ≤ 1.44 g/day
   4. Oral, SC, or IM methotrexate ≤ 25 mg/week
   5. Mizoribine ≤ 150 mg/day (Japan only)
   6. Oral prednisone or equivalent (see Appendix E1) ≤ 40 mg/day
   7. Biologics (eg, belimumab, rituximab).
3. Provided written informed consent before any program-related procedures are performed.
4. Adequate peripheral venous access.
5. Females of childbearing potential must use two effective methods of avoiding pregnancy, only one of which is a barrier method, from screening until 12 weeks after final dose of anifrolumab, unless the patient is surgically sterile (eg, bilateral oophorectomy or complete hysterectomy), has a sterile male partner, is at least 1-year postmenopausal, or practises sustained abstinence consistent with the patient's customary lifestyle. Postmenopausal is defined as at least 1 year since last menses and the patient has an elevated FSH level greater than the local laboratory value of postmenopausal at screening - as detailed in Section 5.4.3.
6. All males (sterilised or non-sterilised) who are sexually active must use a condom (with spermicide where commercially available) from Day 1 (first dose of anifrolumab) until at least 12 weeks after receiving the final dose of anifrolumab. It is strongly recommended that the female partner of a male patient also uses an effective method of contraception (see Section 5.4.3) (other than a barrier method) throughout this period. Male patients must not donate sperm while taking part in the EAP and for 12 weeks after their last dose of anifrolumab - see Section 5.4.3 for further details.
7. Females with an intact cervix must have a documented normal Pap smear without documented malignancy (eg, no signs of CIN grade III, CIS or AIS) within 2 years of entering this EAP and receiving anifrolumab. Any abnormal Pap smear result documented within 2 years before receiving anifrolumb must be repeated to confirm patient eligibility.
8. COVID-19: Any negative PCR test result (central laboratory) at screening and no known or suspected COVID-19 exposure within 2 weeks prior to screening. If there is a known or suspected exposure, a patient must be negative upon retest obtained after 2 weeks and must remain asymptomatic for inclusion in the program. Note: Patients positive at screening may be re-screened after 3 months provided there has been no development of severe COVID-19 disease or sequalae.

Exclusion criteria:

1. Discontinued anifrolumab or placebo before completing Year 3 of the treatment period for study D3461C0009 or study CD1145.
2. Major medical event, such as CVA, MI, malignancy, opportunistic infection, suicide attempt, or that, in the opinion of the Treating Physician, would interfere with patient safety.
3. Any condition that, in the opinion of the Treating Physician, would interfere with patient safety.
4. Active severe or unstable neuropsychiatric SLE where, in the opinion of the Treating Physician, protocol-specified standard therapy is insufficient and utilisation of a more aggressive therapeutic approach, such as adding IV cyclophosphamide and/or high-dose IV pulse corticosteroid therapy or other treatments not permitted in the protocol, is indicated.
5. Active severe SLE-driven renal disease where, in the opinion of the Treating Physician or delegate, protocol-specified standard therapy is insufficient and utilisation of a more aggressive therapeutic approach, such as adding IV cyclophosphamide and/or high-dose IV pulse corticosteroid therapy or other treatments not permitted in the protocol, is indicated.
6. Is receiving any of the following medications:

   1. Azathioprine > 200 mg/day
   2. Mycophenolate mofetil > 2 g/day or mycophenolic acid > 1.44 g/day
   3. Oral, SC, or IM methotrexate > 25 mg/week
   4. Oral prednisone > 40 mg/day (or prednisone equivalent - see Appendix E1)
   5. Mizoribine > 150 mg/day
   6. Biologics eg, belimumab, rituximab
7. Received any of the following:

   1. Live or attenuated vaccine within 8 weeks before signing the ICF. Note: administration of inactivated vaccines is acceptable - the Sponsor recommends that Treating Physicians ensure all patients are up to date on required vaccinations, including influenza (inactivated/recombinant) before EAP entry.
   2. Restricted medications listed in Appendix D if the washout period is not met.
8. Received any investigational product (small molecule or biologic agent) within 4 weeks or 5 half-lives (whichever is greater) before signing the ICF (see Appendix D).
9. Received any commercially available biologic agent within 5 half-lives before signing ICF (see Appendix D).
10. Received B-cell-depleting therapy (including, but not limited to: ocrelizumab, ofatumumab, atacicept, obinutuzumab, rituximab) within 26 weeks before signing the ICF; within 40 weeks for atacicept (see Appendix D) or if therapy was administered 26 weeks or more ago (40 weeks for atacicept), absolute B-cell count should not be less than the LLN or baseline (whichever is lower) before receipt of B-cell-depleting therapy.
11. Positive hepatitis B, hepatitis C or HIV.
12. Known history of allergy or reaction to any component of anifrolumab or history of anaphylaxis to any human gamma globulin therapy.
13. COVID-19: Any history of severe COVID-19 infection (e.g. requiring hospitalisation, ICU care or assisted ventilation) or any prior COVID-19 infection with unresolved sequelae. Any acute COVID-19 infection (laboratory confirmed or suspected based on clinical symptoms) within the last 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult